CLINICAL TRIAL: NCT06522230
Title: Analyzing the Perceived Impact of Fascial Stretch Therapy on the Post-exercise Recovery Process.
Brief Title: Post Exercise Recovery and FST
Acronym: FST
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of British Columbia (Other)
Responsible Party: Principal Investigator, Tanya Forneris, Professor of Teaching, University of British Columbia
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: H24-00681
Record Dates: First submitted 2024-07-10; First posted 2024-07-26 (Actual); Last update posted 2024-08-23 (Actual); Status verified 2024-08

CONDITIONS: Exercise Therapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Fascial Stretch Therapy Intervention (Experimental): Participants receive 3 x 30 Minutes of Fascial Stretch Therapy (FST). FST is designed to enhance flexibility and functional range of motion. During these sessions, participant will be lying down comfortably while a trained therapist gently stretches their body. The therapist will use a mix of pulling, gentle movements, and controlled stretches to loosen up the connective tissue around your muscles and joints.
  Interventions: Other: Fascial Stretch Therapy

INTERVENTIONS:
Other: Fascial Stretch Therapy — Fascial Stretch Protocol uses a combination of circumduction, traction, proprioceptive neuromuscular facilitation (PNF) and specific FST maneuvers. Stretch is applied in both active & passive methods taking into consideration: (1) Oscillatory - slow passive joint oscillations (back and forth movement in a regular rhythm). Small controlled oscillations help with proprioceptors around the joints, acilitates blood flow, gently stretches the ligaments, tendons, nerves, & muscles and slows the nervous system down; (2) Traction - allows for assessment of the joint capsule movement and to decompress the joint. (3) Movement - designed to enhance the reflexes and are intentionally gentle to maximize benefits; (4) PNF - helps improve flexibility by alternating muscle contractions and relaxations. This stimulates the neuromuscular system, allowing muscles to relax deeper and increase range of motion. (5) Breath - allows the body to increase oxygen consumption to facilitate recovery.
  Other Names: FST; Myofascial Stretch Therapy; Assisted Stretch Therapy

SUMMARY:
In this pilot study the focus is to assess the perceived impact of Fascial Stretch Therapy (FST) on post-exercise recovery in University athletes. The objective is to determine if FST can expedite recovery and enhance overall well-being by reducing muscle soreness and fatigue. The FST protocol will be implement by a certified FST level 2 practitioner. Upon completion of the FST intervention athletes will complete a self-assessment questionnaire. The study aims to provide empirical support for FST's efficacy in improving post-exercise recovery and contributing to the health and performance of university athletes.

DETAILED DESCRIPTION:
Purpose: The purpose of this pilot study is to examine the perceived effects of Fascial Stretch Therapy (FST) on post-exercise recovery among university athletes at UBCO. By focusing solely on this aspect, the study aims to provide a nuanced understanding of how FST influences recovery processes in the context of rigorous athletic training.

Hypothesis: We hypothesize that integrating FST into the post-exercise routine of university athletes will result in expedited recovery, manifested through reduced muscle soreness and fatigue. We expect that the tailored FST sessions will contribute positively to the athletes' overall well-being, allowing them to maintain peak performance levels.

Justification: The justification for this study lies in addressing a gap in current research by honing in on the specific impact of FST on post-exercise recovery. As athletes constantly seek methods to optimize their performance, understanding the potential benefits of FST in this context becomes crucial for informed and evidence-based interventions.

Objectives: The primary objective is to assess the efficacy of FST in enhancing post-exercise recovery among university athletes. Specifically, the study aims to analyze the reduction in muscle soreness and fatigue, providing empirical support for the inclusion of FST in athletic recovery programs.

Research Design: This pilot study adopts a mixed methods one group post-test only design to a allow the understanding of perceived FST in enhancing post-exercise recovery. Participants will complete questionnaires and short semi-structured interviews.

Statistical Analysis: This study will employ descriptive statistical analysis for the questionnaire data and thematic analysis for the interview data.

ELIGIBILITY:
Inclusion Criteria:

* Must be an UBCO student athlete who is at least 19 years of age and currently engaged in normal athletic training

Exclusion Criteria:

* Student athletes under 19 years of age or currently have an existing musculoskeletal injury or medical condition preventing you from engaging in normal athletic training.

Ages: 19 Years to 40 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 5 (Estimated)
Dates: Start 2024-09-01 (Estimated); Primary Completion 2025-05-30 (Estimated); Study Completion 2025-06-30 (Estimated)

PRIMARY OUTCOMES:
Perceptions of Fascial Stretch Therapy (FST) on Post-Exercise and Post-Training Recovery Among UBCO Varsity Athletes | Interviews will be conducted within one week after the completion of the 4th FST session.
  This study aims to assess the perceptions of UBCO varsity athletes regarding the impact of Fascial Stretch Therapy (FST) on their post-exercise and post-training recovery. Participants will undergo a 30-minute FST intervention for four sessions over four weeks. Semi-structured interviews will be conducted with participants post-intervention to gain an understanding of their experiences with FST as part of their athletic training and conditioning.

SECONDARY OUTCOMES:
Improvement in overall range of motion and functioning | through study completion, an average of 1 month
  Assessed using the SF-36, a widely used tool for measuring health-related quality of life (HRQoL). All items are scored so that a high score defines a more favorable health state. In addition, each item is scored on a 0 to 100 range so that the lowest and highest possible scores are 0 and 100, respectively. Scores represent the percentage of total possible score achieved.
Improvement in overall range of motion - back | through study completion, an average of 1 month
  Assessed using the Revised Oswestry Disability Index (RODI) which evaluates perceived functional limitations related to lower back pain. Each of the 10 sections is scored separately (0 to 5 points each) and then added up (max total = 50). Higher scores are indicative of greater disability.
Improvement in overall range of motion - neck | through study completion, an average of 1 month
  Assessed using The Neck Disability Index (NDI) questionnaire which assesses perceived functional limitations related to neck pain. Each section is scored on a 0 to 5 rating scale, in which zero means 'No pain' and 5 means 'Worst imaginable pain'.

IPD SHARING:
Plan to Share IPD: No
There is not a plan to make IPD available.

REFERENCES:
- [Background] Batool SA, Shakil-Ul-Rehman S, Tariq Z, Ikram M. Effects of fasciatherapy versus fascial manipulation on pain, range of motion and function in patients with chronic neck pain. BMC Musculoskelet Disord. 2023 Oct 5;24(1):789. doi: 10.1186/s12891-023-06769-0. PMID 37798756
- [Background] Raja G P, Bhat N S, Fernandez-de-Las-Penas C, Gangavelli R, Davis F, Shankar R, Prabhu A. Effectiveness of deep cervical fascial manipulation and yoga postures on pain, function, and oculomotor control in patients with mechanical neck pain: study protocol of a pragmatic, parallel-group, randomized, controlled trial. Trials. 2021 Aug 28;22(1):574. doi: 10.1186/s13063-021-05533-w. PMID 34454582
- [Background] Ruiz JJB, Perez-Cruzado D, Llanes RP. Immediate effects of lumbar fascia stretching on hamstring flexibility: A randomized clinical trial. J Back Musculoskelet Rehabil. 2023;36(3):619-627. doi: 10.3233/BMR-210274. PMID 36872764